CLINICAL TRIAL: NCT05670587
Title: A Multi-center, Longitudinal 12-week Pilot Study to Evaluate Cough Severity and Its Impact, Utilizing a Next Generation Cough Monitor, in Participants With Idiopathic Pulmonary Fibrosis (IPF) or Non IPF Pulmonary Fibrosis
Brief Title: A Study in People With Pulmonary Fibrosis to Monitor Cough With a Wearable Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1490-0005
Record Dates: First submitted 2022-12-15; First posted 2023-01-04 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Pulmonary Fibrosis
MeSH Terms: conditions — Pulmonary Fibrosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Participants with IPF or non IPF pulmonary fibrosis (Experimental): Participants with IPF or non IPF pulmonary fibrosis.
  Interventions: Device: A wearable cough monitoring device, the Strados Labs RESPᵀᴹ sensor, with an accompanying mobile application (App) for data collection

INTERVENTIONS:
Device: A wearable cough monitoring device, the Strados Labs RESPᵀᴹ sensor, with an accompanying mobile application (App) for data collection — A wearable cough monitoring device, the Strados Labs Remote Electronic Stethoscope Platform (RESP)ᵀᴹ sensor, with an accompanying mobile application (App) for data collection.

SUMMARY:
This study is open to adults aged 18 years and older who have pulmonary fibrosis with or without a known cause (or other forms of pulmonary fibrosis).

The purpose of this study is to better understand coughing in people with pulmonary fibrosis. To do this, a wearable cough monitor called Strados Remote Electronic Stethoscope Platform (RESP) is used. This device will measure how often and how forceful coughing is in people with pulmonary fibrosis.

All participants in the study get the device. It is placed on their skin over the chest.

Participants are in the study for 3 months. During this time, they visit the study site 2 to 3 times. 4 visits are done at the participant's home by video call with the site staff.

During the study, the device measures coughing over 24 hours. This is done on 4 days. Participants fill in questionnaires about their coughing and doctors regularly check participant's lung function. A breathing test that measures how well the lungs are working is performed both in the office and during home visits. The doctors also regularly check participants' health and take note of any unwanted effects.

This study will also record patients' experiences using the cough monitor and video assisted breathing tests at visits 3, 4, 5 and 6 at home.

ELIGIBILITY:
Inclusion criteria

* Provision of signed informed consent in writing prior to study data collection
* Subject aged 18 years or over
* Subject diagnosed with Non-Idiopathic Pulmonary Fibrosis (IPF) Pulmonary Fibrosis (>10% fibrosis on High Resolution Computed Tomography (HRCT) by principal investigator assessment) or IPF as per American Thoracic Society/European Respiratory Society/Japanese Respiratory Society/Asociación Latinoamericana de Tórax (ATS/ERS/JRS/ALAT) Guidelines within the past 12 months
* Forced Vital Capacity (FVC) > 40% predicted at baseline visit
* Life expectancy > 6 months (per assessment of treating physician)

Exclusion criteria

* Current smokers
* Upper Respiratory Tract Infection (URI) or Lower Respiratory Tract Infection (LRTI, including Coronavirus Disease (COVID)-19 infection) within 4 weeks of screening visit
* Airflow obstruction (Forced expiratory volume in one second (FEV1)/FVC < 70%) at baseline or known history of significant spirometry response to bronchodilator
* Cough due to etiology other than Interstitial Lung Disease (ILD) (e.g., allergic rhinitis, Gastroesophageal Reflux Disease (GERD))
* Other respiratory disorders including, but not limited to, a current diagnosis of any obstructive disease including chronic obstructive pulmonary disease (COPD) and asthma, active tuberculosis, lung cancer in treatment or in medical history, sleep apnea, known alpha-1 antitrypsin deficiency, cor pulmonale, clinically significant pulmonary hypertension, clinically significant bronchiectasis, or other active pulmonary diseases.
* Initiation or change in dose or type of anti-tussive medication, angiotensin-converting enzyme (ACE) inhibitors, opiates, and systemic or inhaled (excluding intranasal) corticosteroids in the 4 weeks prior to study entry
* Subject with ILD exacerbation as defined by investigators within 4 weeks prior to study entry
* Subject participating in a clinical study of a systemic or inhaled drug at the time of enrollment
* further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2023-01-16 (Actual); Primary Completion 2024-02-22 (Actual); Study Completion 2024-03-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (13):
- United States (4):
  - Critical Care, Pulmonary and Sleep Associates, Lakewood, Colorado
  - Renown Regional Medical Center, Reno, Nevada
  - Southeastern Research Center, Winston-Salem, North Carolina
  - Lowcountry Lung and Critical Care, Charleston, South Carolina
- Belgium (4):
  - Aalst - HOSP Onze-Lieve-Vrouw, Aalst
  - Jessa Ziekenhuis - Campus Virga Jesse, Hasselt
  - Kortrijk - HOSP AZ Groeninge Kennedylaan, Kortrijk
  - Roeselare - HOSP AZ Delta, Roeselare
- Germany (2):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Universitätsklinikum Jena, Jena
- Netherlands (3):
  - Rijnstate Hospital, Arnhem
  - Amphia Ziekenhuis, Breda
  - Erasmus Medisch Centrum, Rotterdam

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization). For more details refer to: https:// www.mystudywindow.com/msw/datatransparency

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-centre, non-randomised, low intervention, 12-week longitudinal pilot trial in patients with idiopathic pulmonary fibrosis (IPF) or non-IPF pulmonary fibrosis to monitor cough with a wearable device.
Pre-assignment Details: Each subject signed and dated an informed consent form (ICF) according to the local regulatory and legal requirements. All subjects were informed that they were free to withdraw their consent at any time during the trial without penalty or prejudice. The subjects were informed that their personal trial related data would be considered confidential and used by Boehringer Ingelheim in accordance with the local data protection laws.
Groups:
- Participants With IPF or Non IPF Pulmonary Fibrosis: Participants with idiopathic pulmonary fibrosis (IPF) or non IPF pulmonary fibrosis. The Strados Remote Electronic Stethoscope Platform (RESP™) Wearable Cough Monitor, adhered to chest wall, was worn for 24 hours.
Period: Overall Study
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Started | 53
Completed (Completed planned observation period) | 50
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Population: Entered Set (ES): All subjects entered into the study.
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 53
Age, Continuous [Mean (Standard Deviation); unit: Years] | 70.4 (8.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 38
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 53
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 50
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Cough Count Per Hour (CC/hr) Measured Over a 24-hour Period at Baseline Visit, Week 4, Week 8, and at Day 82
Description: Cough count per hour (CC/hr) measured over a 24-hour period at baseline visit, Week 4, Week 8, and at Day 82.
Time Frame: At baseline (Visit 2), Week 4 (Visit 4), Week 8 (Visit 5) and at Day 82 (Visit 6).
Population: Entered Set (ES): All subjects entered into the study. Only participants with non-missing data at the respective timepoints were included in the analysis.
Measure: Mean (Standard Deviation); unit: Cough count per hour
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 53
Cough count per hour
  Baseline: number analyzed (Participants) | 52
  Baseline | 10.79 (14.57)
  Week 4: number analyzed (Participants) | 45
  Week 4 | 12.63 (19.02)
  Week 8: number analyzed (Participants) | 44
  Week 8 | 10.36 (18.03)
  Day 82: number analyzed (Participants) | 39
  Day 82 | 12.45 (17.15)

2. Secondary Outcome: Change From Baseline (CfB) in Cough Count Per Hour (CC/h) at Week 4, Week 8 and at Day 82
Description: Change from baseline (CfB) in cough count per hour (CC/h) at Week 4, Week 8 and at Day 82. Cough count per hour (CC/h) was measured over a 24-h period.
Time Frame: At baseline (Visit 2), Week 4, (Visit 4) Week 8 (Visit 5) and at Day 82 (Visit 6).
Population: Entered Set (ES): All subjects who entered into the study. Only participants with non-missing values at the respective timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: Cough count per hour
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 53
Cough count per hour
  CfB at Week 4: number analyzed (Participants) | 45
  CfB at Week 4 | 1.42 (9.67)
  CfB at Week 8: number analyzed (Participants) | 44
  CfB at Week 8 | 0.12 (8.82)
  CfB at Day 82: number analyzed (Participants) | 39
  CfB at Day 82 | 1.03 (9.01)
Statistical Analysis 1: Comparison: Participants With IPF or Non IPF Pulmonary Fibrosis; Geometric mean (gMean) ratio of change from baseline (CfB) in cough count per hour (CC/h) at Week 4; Test type: Other; gMean ratio at Week 4 = 0.95, 95% CI 2-sided [0.76 to 1.18] — gMean ratios of CfB in CC/h were calculated from the log transformed values at each visit. Geometric Coefficient of variation (gCV) = 84.59%
Statistical Analysis 2: Comparison: Participants With IPF or Non IPF Pulmonary Fibrosis; Geometric mean (gMean) ratio of change from baseline (CfB) in cough count per hour (CC/h) at Week 8; Test type: Other; gMean ratio at Week 8 = 0.84, 95% CI 2-sided [0.64 to 1.11] — gMean ratios of CfB in CC/h were calculated from the log transformed values at each visit. Geometric coefficient of variation (gCV) = 115.62%
Statistical Analysis 3: Comparison: Participants With IPF or Non IPF Pulmonary Fibrosis; Geometric mean (gMean) ratio of change from baseline (CfB) in cough count per hour (CC/h) at Day 82; Test type: Other; gMean ratio at Day 82 = 0.98, 95% CI 2-sided [0.75 to 1.29] — gMean ratios of CfB in CC/h were calculated from the log transformed values at each visit. Geometric coefficient of variation (gCV) = 100.02%

3. Secondary Outcome: Forced Vital Capacity (FVC) at Baseline and at Week 12
Description: Forced Vital Capacity (FVC) at baseline and at Week 12.
Time Frame: At baseline (Visit 2) and at Week 12 (Visit 7).
Population: Entered Set (ES): All subjects entered into the study. Only participants with non-missing data at the respective timepoint were included in the analysis.
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 53
Milliliter (mL)
  Baseline: number analyzed (Participants) | 52
  Baseline | 3073.8 (881.6)
  Week 12: number analyzed (Participants) | 50
  Week 12 | 3021.1 (869.3)

4. Secondary Outcome: Change From Baseline in Forced Vital Capacity (FVC) at Week 12
Description: Change from baseline in Forced Vital Capacity (FVC) at Week 12.
Time Frame: At baseline (Visit 2) and at Week 12 (Visit 7).
Population: Entered Set (ES): All subjects entered into the study. Only participants with non-missing data were included in the analysis.
Measure: Mean (Standard Deviation); unit: Milliliter (mL)
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 49
Milliliter (mL) | -23.9 (388.2)

5. Secondary Outcome: Percentage (%) of Analysable Cough Device Data Per 24-hour Recording (Feasibility of Remote Cough Data Capture)
Description: Feasibility of remote cough data capture , defined as % of analysable cough device data per 24-hours recording.
  The percentage of analysable data per 24-hours recording period was derived from cough count (CC) recording times (total readable recording time) and defined as:
  (Total readable recording time/24 hours)·100 Percent of analysable cough data is percentage of 24 hours of total expected recording time that was readable.
Time Frame: At baseline (Visit 2), Week 4 (Visit 4), Week 8 (Visit 5) and at Day 82 (Visit 6).
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Percentage (%)
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 53
Percentage (%)
  Baseline: number analyzed (Participants) | 52
  Baseline | 92.0 (20.6)
  Week 4: number analyzed (Participants) | 45
  Week 4 | 93.6 (19.9)
  Week 8: number analyzed (Participants) | 44
  Week 8 | 82.2 (32.2)
  Day 82: number analyzed (Participants) | 39
  Day 82 | 93.1 (18.1)

6. Secondary Outcome: Number of Successful Completion of All Elements of Remote Visit (Feasibility of Hybrid Study Design)
Description: Successful completion of all elements of remote visit (feasibility of hybrid study design). Successful completion of a remote visit was based on the questions on the home trial procedures:
  * Was home spirometry performed?
  * Was the video conference tele-visit completed?
  * Was the 24-hour cough recording completed? The number (percentage) of participants who completed each element is reported by visit.
Time Frame: At Day 3 (Visit 3), Week 4 (Visit 4), Week 8 (Visit 5) and at Day 82 (Visit 6).
Population: Entered Set: All subjects entered into the study. Only participants with non-missing data at the respective timepoint were included in the analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
Number analyzed (Participants) | 51
Participants
  Successful completion on Day 3 | 34
  Successful completion on Week 4 | 36
  Successful completion on Week 8 | 33
  Successful completion on Day 82 | 31

ADVERSE EVENTS:
Time Frame: All-cause mortality, serious and other adverse events: From study start until the individual subject's end of trial visit (V7), up to 12 weeks and 5 days.
Description: Entered Set (ES): All subjects entered into the study.
Arm/Group | Participants With IPF or Non IPF Pulmonary Fibrosis
All-Cause Mortality (participants affected / at risk) | 0/53
Serious Adverse Events (participants affected / at risk) | 0/53
Other Adverse Events (participants affected / at risk) | 0/53

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-09-16): https://cdn.clinicaltrials.gov/large-docs/87/NCT05670587/Prot_000.pdf
  • Statistical Analysis Plan (2024-04-09): https://cdn.clinicaltrials.gov/large-docs/87/NCT05670587/SAP_001.pdf